CLINICAL TRIAL: NCT07093788
Title: Super High-pressure Balloon Versus Intravascular Lithotripsy to Prepare Severely Calcified Coronary Lesions: a Randomized Controlled Trial (Shape)
Brief Title: Super High-pressure Balloon Versus Intravascular Lithotripsy to Prepare Severely Calcified Coronary Lesions
Acronym: Shape
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ye-fei, chief physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20250425-03
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: PCI; Coronary Arterial Disease (CAD); Calcified Coronary Lesions
Keywords: super high-pressure balloon; percutaneous coronary intervention; intravascular lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super high-pressure balloon (Experimental): Patients underwent OCT-guided PCI were treated with super high-pressure balloon for lesion preparation.
  Interventions: Device: super high-pressure balloon
- Intravascular lithotripsy (IVL) (Experimental): Patients underwent OCT-guided PCI were treated with Intravascular lithotripsy (IVL) for lesion preparation.
  Interventions: Device: intravascular lithotripsy (IVL)

INTERVENTIONS:
Device: super high-pressure balloon — preparation strategy for calcified lesions after unsatisfactory dilation
  Arms: Super high-pressure balloon
Device: intravascular lithotripsy (IVL) — preparation strategy for calcified lesions after unsatisfactory dilation
  Arms: Intravascular lithotripsy (IVL)

SUMMARY:
this trial aimed to evaluate the stent expansion through optical coherence tomography (OCT) among individuals underwent different preparation techniques ,then comparing the efficacy and safety of super high-pressure balloon to IVL in severely calcified lesions

DETAILED DESCRIPTION:
Calcified lesions posed a significant challenge in percutaneous coronary intervention (PCI). The existence of calcified plaque increased the difficulty of optimal stent expansion and the risk of target lesion failure(TLF). Consequently, optimizing the preparation techniques for calcified lesions before stent implantation has assumed growing importance.

As a kind of novel double-layered balloon, super high-pressure balloon can expand uniformly under extreme pressure. Previous studies have demonstrated that super high-pressure balloon perform non-inferiorly or superiorly to other strategies in terms of final stent expansion.

Through triggering localized pulsatile sonic pressure, intravascular lithotripsy(IVL) cracked intimal and medial calcium plaque within the artery. In present series of studies(DISRUPT), the optimized preparation of calcified lesions with IVL has been proved to be safe and effective. According to guidelines and clinical practice, IVL is applicable to different types of severe calcification lesions, including concentric and eccentric calcifications. However, considering its technological and economic costs, finding other preparation techniques non-inferiority to IVL was essential. In clinical practice, super high-pressure balloon had shown considerable effects of preparation for calcified lesions. However, study focused on the comparison of super high-pressure balloon with IVL for severe calcified lesions was limited.

In summary, this randomized trial aimed to evaluate the stent expansion through optical coherence tomography (OCT) among individuals underwent different preparation techniques ,then comparing the efficacy and safety of super high-pressure balloon to IVL in severely calcified lesions

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 80 years
* Presented as asymptomatic angina, stable angina, unstable angina, prior myocardial infarction (MI), or non-ST-elevation myocardial infarction (NSTEMI).
* Have an indication for drug-eluting stent (DES) implantation
* Denovo coronary artery calcified lesions
* Target lesion diameter stenosis ≥ 70%, or target lesion diameter stenosis between ≥ 50% and < 70%, accompanied by evidence of myocardial ischemia(such as fractional flow reserve (FFR) ≤ 0.80 or minimal lumen area (MLA) ≤ 4.0 mm²).
* Reference vessel diameter of the target vessel between 2.5 mm - 4.5 mm
* Maximum calcium arc within the lesion ≥ 270⁰ assessed by optical coherence tomography (OCT)
* Unsatisfactory lesion preparation with non-compliant balloon, defined as baseline diameter stenosis reduction of < 30% under maximal inflation pressure.
* Provision of written informed consent

Exclusion Criteria:

* Presented as acute ST-segment elevation myocardial infarction (STEMI), cardiogenic shock and multiple organ failure
* Presented as severe contrast agent allergy
* Intolerant to dual antiplatelet therapy (DAPT) and/or anticoagulation therapy
* Presented as active phase of autoimmune disease
* Calcified nodules or eccentric calcification lesions
* Failure to reach the target lesion with guidewires or catheters
* Complex coronary bifurcation lesions
* Target vessel thrombosis or aneurysm within 10 mm of the target lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
stent expansion index | Intraprocedural
  The stent expansion was associated with post-PCI clinical outcomes and the risk of stent failure.In this study, the primary endpoint was stent expansion index, which was defined as the final minimal luminal area (MLA) within the treated segment divided by the average reference vessel area assessed with optical coherence tomography(OCT).

SECONDARY OUTCOMES:
30-days major adverse cardiac event (MACE) | 30 days
  The secondary endpoint was defined as the occurrence of major adverse cardiac events within 30 days, which was defined as a composite of cardiac death, target vessel-related myocardial infarction [TVMI] and clinically driven target vessel revascularisation[TVR].

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (3):
- China (3):
  - Lianyungang First People's Hospital, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Yixing People's Hospital, Yixing, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Due to privacy and ethical limitations, the data generated and analyzed in current study are not publicly available but could be obtained from principal investigator upon the approval of ethics committee

REFERENCES:
- [Background] Cassese S, Simonetti F, Covarrubias HAA, Janisch M, Joner M, Kufner S, Lenz T, Pellegrini C, Rheude T, Sager H, Schunkert H, Starnecker F, Voll F, Xhepa E, Kastrati A, Kessler T. Intracoronary stenting and additional results achieved by shockWAVE coronary lithotripsy: design and rationale of ISAR-WAVE trial. Am Heart J. 2025 Apr;282:1-12. doi: 10.1016/j.ahj.2024.12.008. Epub 2024 Dec 20. PMID 39710352
- [Background] Sagris M, Ktenopoulos N, Dimitriadis K, Papanikolaou A, Tzoumas A, Terentes-Printzios D, Synetos A, Soulaidopoulos S, Lichtenberg M, Korosoglou G, Honton B, Tousoulis D, Tsioufis C, Toutouzas K. Efficacy of intravascular lithotripsy (IVL) in coronary stenosis with severe calcification: A multicenter systematic review and meta-analysis. Catheter Cardiovasc Interv. 2024 Apr;103(5):710-721. doi: 10.1002/ccd.31006. Epub 2024 Mar 14. PMID 38482928
- [Background] Rheude T, Rai H, Richardt G, Allali A, Abdel-Wahab M, Sulimov DS, Mashayekhi K, Ayoub M, Cuculi F, Bossard M, Kufner S, Xhepa E, Kastrati A, Fusaro M, Joner M, Byrne RA, Cassese S. Super high-pressure balloon versus scoring balloon to prepare severely calcified coronary lesions: the ISAR-CALC randomised trial. EuroIntervention. 2021 Aug 27;17(6):481-488. doi: 10.4244/EIJ-D-20-01000. PMID 33258774
- [Background] Rheude T, Fitzgerald S, Allali A, Mashayekhi K, Gori T, Cuculi F, Kufner S, Hemetsberger R, Sulimov DS, Rai H, Ayoub M, Bossard M, Xhepa E, Fusaro M, Toelg R, Joner M, Byrne RA, Richardt G, Kastrati A, Cassese S, Abdel-Wahab M. Rotational Atherectomy or Balloon-Based Techniques to Prepare Severely Calcified Coronary Lesions. JACC Cardiovasc Interv. 2022 Sep 26;15(18):1864-1874. doi: 10.1016/j.jcin.2022.07.034. PMID 36137691